CLINICAL TRIAL: NCT00774709
Title: Ancillary Study of the Registry Karolinska-Rennes (KaRen) : Prospective Study of Dyssynchrony in Heart Failure With Preserved Ejection Fraction
Brief Title: Karolinska-Rennes (KaRen) Prospective Study of Exercise Stress Echocardiography in Heart Failure With Preserved Ejection Fraction
Acronym: KaRen
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Collaborators: Fédération Française de Cardiologie (Other)
Responsible Party: Sponsor
Other Study IDs: CCP 08 / 20- 679
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Heart Failure
Keywords: Heart failure; Preserved ejection fraction; Diastolic dysfunction; Dyssynchrony; Echocardiography; Patients with acute heart failure clinically; diagnosed; BNP level > 100 ng / l or NT-proBNP > 300 ng /l; Preserved left ventricular ejection fraction(LVEF; ≥ 45%)
MeSH Terms: conditions — Heart Failure; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
Background:

Heart failure with preserved ejection fraction (HFPEF) is common but not well understood. Electrical dyssynchrony in systolic heart failure is harmful. Little is known about the prevalence and the prognostic impact of dyssynchrony in HFPEF.

Methods:

We have designed a prospective, multicentre, international, observational study to characterize HFPEF and to determine whether electrical or mechanical dyssynchrony affects prognosis. Patients presenting with acute heart failure will be screened.

Inclusion criteria will be:

acute presentation with Framingham criteria for heart failure, left ventricular EF ≥45%, BNP >100 ng/L or NT-proBNP >300 ng/L. Patients will return in stable condition 4-8 weeks after the index presentation and undergo questionnaires, serology, ECG and Dopplerechocardiography. Thereafter, patients will be followed for mortality and heart failure hospitalization every 6 months for at least 18 months. Sub-studies will focus on echocardiographic changes from the acute presentation to the stable condition and on exercise echocardiography.

Conclusion:

KaRen aims to characterize electrical and mechanical dyssynchrony and to assess its prognostic impact in the HFPEF. The ancillary study of the exercise stress echocardiography sought to improve our understanding of HFPEF and generate answers to the question whether dyssynchrony could be a target for therapy in HFPEF.

ELIGIBILITY:
Inclusion Criteria:

1. Acute presentation to the hospital with clinical signs and symptoms of HF, according to the Framingham criteria [19].
2. LVEF ≥ 45% by echocardiography within the first 72 hours. The measurement will be carried out according to guidelines
3. BNP >100 ng/L or NT-proBNP >300 ng/L.

Exclusion Criteria:

1. Evidence of primary hypertrophic or restrictive cardiomyopathy or systemic illness known to be associated with infiltrative heart disease
2. Known cause of right heart failure not related to left ventricular dysfunction
3. Pericardial constriction
4. Clinically significant pulmonary disease, as evidenced by requirement of current home oxygen
5. End-stage renal disease currently requiring dialysis
6. Bi-ventricular pacemaker (CRT). (Patients who have a conventional pacemaker may be included)
7. Anticipated or indication for cardiac surgery. (Patients who have indication for surgery but may not undergo surgery because of some contraindication, for example age, may NOT be included).
8. Anticipated percutaneous intervention on aortic stenosis. (Patients who undergo other percutaneous intervention, for example PCI, may be included).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting acutely of congestive heart failure and diagnosed according to current ESC guidelines to have an heart failure with preserved ejection fraction (LV EF > or = 45%)
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Echocardiographic parameter | 4 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erwan Donal, MD, PhD, Principal Investigator — Service de Cardiologie - CHU Rennes
Locations (1):
- Service de Cardiologie et CIT-IC 804, LTSI INSERM U 642, Rennes, France

REFERENCES:
- [Derived] Lund LH, Savarese G, Venkateshvaran A, Benson L, Lundberg A, Donal E, Daubert JC, Oger E, Linde C, Hage C. Eligibility of patients with heart failure with preserved ejection fraction for sacubitril/valsartan according to the PARAGON-HF trial. ESC Heart Fail. 2022 Feb;9(1):164-177. doi: 10.1002/ehf2.13705. Epub 2021 Nov 22. PMID 34811954
- [Derived] Hage C, Wardell E, Linde C, Donal E, Lam CSP, Daubert C, Lund LH, Mansson-Broberg A. Circulating neuregulin1-beta in heart failure with preserved and reduced left ventricular ejection fraction. ESC Heart Fail. 2020 Apr;7(2):445-455. doi: 10.1002/ehf2.12615. Epub 2020 Jan 24. PMID 31981321
- [Derived] Hage C, Bjerre M, Frystyk J, Gu HF, Brismar K, Donal E, Daubert JC, Linde C, Lund LH. Comparison of Prognostic Usefulness of Serum Insulin-Like Growth Factor-Binding Protein 7 in Patients With Heart Failure and Preserved Versus Reduced Left Ventricular Ejection Fraction. Am J Cardiol. 2018 Jun 15;121(12):1558-1566. doi: 10.1016/j.amjcard.2018.02.041. Epub 2018 Mar 14. PMID 29622288
- [Derived] Nagy AI, Hage C, Merkely B, Donal E, Daubert JC, Linde C, Lund LH, Manouras A. Left atrial rather than left ventricular impaired mechanics are associated with the pro-fibrotic ST2 marker and outcomes in heart failure with preserved ejection fraction. J Intern Med. 2018 Apr;283(4):380-391. doi: 10.1111/joim.12723. Epub 2018 Feb 12. PMID 29430747
- [Derived] Donal E, Lund LH, Oger E, Bosseau C, Reynaud A, Hage C, Drouet E, Daubert JC, Linde C; KaRen Investigators. Importance of combined left atrial size and estimated pulmonary pressure for clinical outcome in patients presenting with heart failure with preserved ejection fraction. Eur Heart J Cardiovasc Imaging. 2017 Jun 1;18(6):629-635. doi: 10.1093/ehjci/jex005. PMID 28329385
- [Derived] Hage C, Michaelsson E, Linde C, Donal E, Daubert JC, Gan LM, Lund LH. Inflammatory Biomarkers Predict Heart Failure Severity and Prognosis in Patients With Heart Failure With Preserved Ejection Fraction: A Holistic Proteomic Approach. Circ Cardiovasc Genet. 2017 Feb;10(1):e001633. doi: 10.1161/CIRCGENETICS.116.001633. PMID 28100627
- [Derived] Bosseau C, Donal E, Lund LH, Oger E, Hage C, Mulak G, Daubert JC, Linde C; KaRen investigators. The prognostic significance of atrial fibrillation in heart failure with preserved ejection function: insights from KaRen, a prospective and multicenter study. Heart Vessels. 2017 Jun;32(6):735-749. doi: 10.1007/s00380-016-0933-8. Epub 2016 Dec 27. PMID 28028584
- [Derived] Hage C, Lund LH, Donal E, Daubert JC, Linde C, Mellbin L. Copeptin in patients with heart failure and preserved ejection fraction: a report from the prospective KaRen-study. Open Heart. 2015 Nov 3;2(1):e000260. doi: 10.1136/openhrt-2015-000260. eCollection 2015. PMID 26568833
- [Derived] Donal E, Lund LH, Oger E, Hage C, Persson H, Reynaud A, Ennezat PV, Bauer F, Sportouch-Dukhan C, Drouet E, Daubert JC, Linde C; KaRen Investigators. Baseline characteristics of patients with heart failure and preserved ejection fraction included in the Karolinska Rennes (KaRen) study. Arch Cardiovasc Dis. 2014 Feb;107(2):112-21. doi: 10.1016/j.acvd.2013.11.002. Epub 2013 Dec 30. PMID 24388161